CLINICAL TRIAL: NCT04894877
Title: International Study of Comparative Health Effectiveness With Medical and Invasive Approaches (ISCHEMIA) Extended Follow-up
Brief Title: ISCHEMIA-EXTEND (Extended Follow-up)
Status: Active, not recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: New York University (Other); Stanford University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: 11-00498-2; 1R01HL149888 (NIH)
Record Dates: First submitted 2021-05-18; First posted 2021-05-20 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Coronary Artery Disease; Heart Diseases; Myocardial Ischemia
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Coronary Artery Disease; Heart Diseases; Myocardial Ischemia | interventions — Cardiac Catheterization; Coronary Artery Bypass; Percutaneous Coronary Intervention; Dosage Forms; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active Comparator: Invasive Strategy (INV): Routine invasive strategy with cardiac catheterization followed by revascularization plus optimal medical therapy.
  Interventions: Procedure: cardiac catheterization; Procedure: coronary artery bypass graft surgery; Procedure: percutaneous coronary intervention
- Active Comparator: Conservative Strategy: Optimal medical therapy with cardiac catheterization and revascularization reserved for patients with acute coronary syndrome, ischemic heart failure, resuscitated cardiac arrest or refractory symptoms.
  Interventions: Behavioral: Lifestyle; Drug: Medication

INTERVENTIONS:
Procedure: cardiac catheterization — Narrowed blood vessels can be opened without surgery using stents or can be bypassed with surgery. To determine which is the best approach for you the doctor needs to look at your blood vessels to see where the narrowings are and how much narrowing there is. This is done by a procedure known as a cardiac catheterization.
  Other Names: Cath
  Groups: Active Comparator: Invasive Strategy (INV)
Procedure: coronary artery bypass graft surgery — Artery narrowing is bypassed during surgery with a healthy artery or vein from another part of the body. This is known as coronary artery bypass grafting, or CABG (said, "cabbage"). The surgery creates new routes around narrowed and blocked heart arteries. This allows more blood flow to the heart.
  Other Names: CABG
  Groups: Active Comparator: Invasive Strategy (INV)
Procedure: percutaneous coronary intervention — Percutaneous coronary intervention may be done as part of the cardiac catheterization procedure. With this procedure a small, hollow, mesh tube (stent) is inserted into the narrowed part of the artery. The stent pushes the plaque against the artery wall, and opens the vessel to allow better blood flow.
  Other Names: PCI
  Groups: Active Comparator: Invasive Strategy (INV)
Behavioral: Lifestyle — diet, physical activity, smoking cessation
  Other Names: Behavior change
  Groups: Active Comparator: Conservative Strategy
Drug: Medication — antiplatelet, statin, other lipid lowering, antihypertensive, and anti-ischemic medical therapies
  Other Names: Pharmacologic Therapy
  Groups: Active Comparator: Conservative Strategy

SUMMARY:
The International Study of Comparative Health Effectiveness with Medical and Invasive Approaches (ISCHEMIA) Extended Follow-up (ISCHEMIA-EXTEND) is the long-term follow-up of randomized, surviving participants in ISCHEMIA. ISCHEMIA was an NHLBI-supported trial that randomized 5,179 participants with stable ischemic heart disease to two different management strategies: 1) an initial invasive strategy (INV) of cardiac catheterization and revascularization when feasible plus guideline-directed medical therapy (GDMT), or 2) an initial conservative strategy (CON) of GDMT. The trial did not demonstrate a reduction in the primary endpoint with an initial invasive strategy. There was an excess of procedural myocardial infarction (MI) and a reduction in spontaneous MI in the INV group. Prior evidence suggests that spontaneous MI carries a higher risk of subsequent death than procedural MI. There was a late separation in the cardiovascular (CV) mortality curves over a median of 3.2 years follow-up in ISCHEMIA. The MI incidence curves crossed at approximately 2 years. However, during the trial follow-up phase there were excess non-CV deaths in the invasive strategy. Therefore, it is imperative to ascertain long-term vital status to provide patients and clinicians with robust evidence on whether there are differences between management strategies and to increase precision around the treatment effect estimates for risk of all-cause, CV and non-CV death over the long-term.

Overarching Goal:

To assess the effect of an initial invasive strategy on long-term all-cause, CV and non-CV mortality compared with an initial conservative strategy in SIHD patients with at least moderate ischemia on stress testing, over 10 years median follow-up.

Condition: Coronary Disease Procedure: Observational Phase: Phase III per NIH Condition: Cardiovascular Diseases Procedure: Observational Phase: Phase III per NIH Condition: Heart Diseases Procedure: Observational Phase: Phase III per NIH

DETAILED DESCRIPTION:
The primary goals of all therapies are to enable patients to feel better and/or live longer. ISCHEMIA provided definitive data on the benefit of INV on quality of life. However, mortality is the most objective and compelling clinical outcome. Strategies that reduce deaths over the long term are of greatest interest to patients and physicians. Long-term follow-up of the ISCHEMIA trial cohort to assess all-cause, CV and non-CV mortality by treatment group is particularly important given that the primary results show relatively late crossing of the event curves, an overall reduction in spontaneous MI with INV, and late divergence of CV death curves in favor of the INV strategy but with an excess of non-CV deaths.

DESIGN NARRATIVE, INCLUDING MODIFICATIONS DURING THE TRIAL:

The investigators will conduct a long-term ascertainment of all-cause, CV and non-CV mortality for surviving ISCHEMIA participants. The limited follow-up after the observed reduction in spontaneous MI events may not have been long enough to observe a mortality benefit, and this makes it imperative to assess long-term all-cause, CV and non-CV mortality to determine whether an initial invasive strategy reduces the risk of death years later, as seen in other trials with crossing curves, e.g., STICH, a randomized trial comparing a strategy of surgical revascularization to GDMT alone in patients with SIHD and LVEF <35%.

Furthermore, with additional accrual of deaths, the investigators will provide estimates on the impact of INV in the highest risk subgroup, those with coronary artery anatomy for whom practice guidelines have recommended CABG to improve survival (3-vessel CAD and 2-vessel CAD with proximal LAD stenosis). Equally important is to improve precision around the point estimates of the treatment effect for all-cause, CV and non-CV mortality for the trial overall and in important subgroups to efficiently maximize the substantial investment by of NHLBI, patients, and study teams.

Vital status data will be collected in a rigorous manner from high-quality vital statistics registries, medical records, or by contacting participants and their next of kin.

ISCHEMIA-EXTEND will also follow eligible participants from the NHLBI-funded ISCHEMIA-CKD trial with the same methodology as for the main trial with separate analyses. They will be referred to as ISCHEMIA-EXTEND for the main trial and ISCHEMIA-CKD EXTEND for the CKD trial.

PARTICIPATING COUNTRIES:

North America: Canada; Mexico; USA South America: Argentina; Brazil; Peru Asia: China; India; Japan; Malaysia; Singapore; Thailand; Russian Federation Pacifica: Australia; New Zealand Europe: Austria; Belgium; France; Germany; Hungary; Italy; Lithuania; Macedonia; Netherlands; Poland; Portugal; Romania; Serbia; Spain; Sweden; Switzerland; UK Middle East: Egypt; Israel; Saudi Arabia Africa: South Africa

ELIGIBILITY:
Inclusion Criteria:

* Alive at the end of the initial follow-up period for ISCHEMIA

Exclusion Criteria:

* Participants who withdrew consent during initial trial phase
* Participants who declined participation in long-term follow-up

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants of the ISCHEMIA main trial that meet the EXTEND inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 5391 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative Event Rate of Death: All-Cause | Year 10 (Range: 6-13 years)
  Cumulative event rate of death from all causes.
Cumulative Event Rate of Cardiovascular (CV) Death | Year 10 (Range 6-13 years)
  Cumulative event rate of death from cardiovascular causes.
Cumulative Event Rate of Non-CV Death | Year 10 (Range: 6-13 years)
  Cumulative event rate of death from non-cardiovascular causes.

SECONDARY OUTCOMES:
Cumulative Event Rate of Death by High Risk Subgroups | Year 10 (Range 6-13 years)
  Angiographic and clinical risk variables.

CONTACTS AND LOCATIONS:
Overall Officials: Judith S Hochman, MD, Principal Investigator — New York University

IPD SHARING:
Plan to Share IPD: Yes
Data from the follow-up analysis will be made available 2 years after the main results paper is published.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article
URL: http://www.ischemiatrial.org/

REFERENCES:
- [Derived] Hochman JS, Anthopolos R, Reynolds HR, Bangalore S, Xu Y, O'Brien SM, Mavromichalis S, Chang M, Contreras A, Rosenberg Y, Kirby R, Bhargava B, Senior R, Banfield A, Goodman SG, Lopes RD, Pracon R, Lopez-Sendon J, Maggioni AP, Newman JD, Berger JS, Sidhu MS, White HD, Troxel AB, Harrington RA, Boden WE, Stone GW, Mark DB, Spertus JA, Maron DJ; ISCHEMIA-EXTEND Research Group. Survival After Invasive or Conservative Management of Stable Coronary Disease. Circulation. 2023 Jan 3;147(1):8-19. doi: 10.1161/CIRCULATIONAHA.122.062714. Epub 2022 Nov 6. PMID 36335918

DOCUMENTS (1):
  • Study Protocol (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT04894877/Prot_000.pdf